CLINICAL TRIAL: NCT01601561
Title: The Effect of Insulin on Protein Metabolism After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09-105-SDR
Record Dates: First submitted 2012-03-09; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Cardiac Surgery
Keywords: Insulin; Protein metabolism; Stress response
MeSH Terms: conditions — Insulin Resistance; Fractures, Stress | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-dose insulin (Experimental)
  Interventions: Drug: Regular human insulin injection
- Control (No Intervention)

INTERVENTIONS:
Drug: Regular human insulin injection — Hyperinsulinemic normoglycemic clamp from beginning of surgery until 8 hours after surgery.
  Humulin R 5 mU/kg/min and a variable infusion of glucose.
  Other Names: Humulin R
  Arms: High-dose insulin

SUMMARY:
Background: The hyperinsulinemic-normoglycaemic clamp technique is a precise method of providing insulin and glucose while maintaining normoglycemia. High-dose insulin has profound effects on glucose and protein metabolism. It has been demonstrated in coronary artery bypass graft (CABG) surgery patients that high-dose insulin causes hypoaminoacidaemia. The investigators hypothesize that the reduction of plasma amino acids (AAs) levels as seen in patients undergoing CABG surgery and receiving high-dose insulin is a consequence of an inhibition of whole body proteolysis as assessed by L-[1-13C]leucine tracer kinetics.

Objective: The present study aims to investigate the effect of high-dose insulin therapy on whole body protein, glucose and end-organ metabolism in patients undergoing CABG surgery using stable isotope tracers [6,6-2H2]glucose, L-[1-13C]-leucine and L-[2H5]phenylalanine. The changes in the metabolic-endocrine milieu will also be evaluated by plasma concentrations of glucose, lactate, free fatty acids, prealbumin, albumin, fibrinogen, insulin, glucagon, and cortisol.

Methods: With the approval of local institution's ethical committee, 30 patients scheduled for elective will be enrolled. The patients will be divided randomly into two groups. The control group will receive a standard IV insulin protocol with the aim of keeping blood glucose < 10 mmol/L. The treatment group will be administered a high dose insulin infusion of 5 mU/kg/min coupled with a variable infusion of glucose to maintain normoglycemia (4-6 mmol/L). Insulin infusion will be continued until the end of the study period approximately 8 hours after surgery. L-[1-13C]leucine and [6,6-2H2]glucose kinetics will be used to assess changes in whole body protein and glucose kinetics. Hepatic albumin synthesis will be determined by using primed continuous infusion of L-[2H5]phenylalanine. The preoperative measurements will be performed on the morning before the surgery. Postoperative studies will be conducted two hours after arrival in the intensive care unit. Tracer kinetics between the two groups will be analyzed using ANOVA for repeated measurements.

Significance: High-dose-insulin results in a significant reduction in plasma AAs in cardiac surgery. This study should address if this drop in plasma AA levels is secondary to a decrease in breakdown, an increase in synthesis or both during high-dose insulin therapy in open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent

Exclusion Criteria:

* signs of severe malnutrition or obesity: body mass index (BMI) < 20 or > 30 kg.m-2, more than 10% involuntary body weight loss over the preceding six months, serum albumin < 35 g.L-1
* chronic liver failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Protein breakdown | Eight hours after the end of surgery
  Protein breakdown as measured by 13C leucine

CONTACTS AND LOCATIONS:
Overall Officials: Roupen Hatzakorzian, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, McGill University Health Centre, Montreal, Quebec, Canada